CLINICAL TRIAL: NCT07058142
Title: The Effects of an Interaction Standard Theory-Based Multi-Care Program on Postpartum Recovery, Coping Styles, Psychological Distress, and Quality of Life in Women With Postpartum Hemorrhage
Brief Title: Effects of an Interaction-Based Multi-Care Program on Postpartum Hemorrhage Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xingxing Lv (Other)
Responsible Party: Sponsor-Investigator, Xingxing Lv, Principal Investigator, Shijiazhuang Obstetrics and Gynecology Hospital
Organization: Shijiazhuang Obstetrics and Gynecology Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-SOG-23
Record Dates: First submitted 2025-06-24; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Hemorrhage; Postpartum Period; Psychological Distress; Quality of Life
Keywords: Interaction standard theory-based multi-care; Postpartum hemorrhage; Postpartum recovery; Quality of life; Coping styles; Psychological distress; Nursing intervention
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interaction Standard Theory-Based Multi-Care Program Group (Experimental): Participants received conventional nursing care plus an interaction standard theory-based multi-care program. This program involved:
  * Collective training for nursing staff on interaction theories and PPH care.
  * One-on-one communication to assess patient's psychological state, background, and needs.
  * Collaborative development of a multi-dimensional care plan.
  * Specific interventions including:
  * Hemorrhage Care: Encouraging early breastfeeding, monitoring bleeding, administering uterotonics if needed, abdominal massage.
  * Psychological Care: Empathetic listening, Satir's communication stances, music therapy, deep breathing, guided imagery.
  * Cognitive Intervention: Education on PPH causes, treatments, complications using various materials.
  * Dietary Care: Scientific, balanced dietary plan emphasizing high-calorie, high-protein foods.
  * Rehabilitation Training: Ensuring warmth, sleep, abdominal massage, gentle vaginal pressure, early ambulation, specific exercises.
  * Implementation
  Interventions: Behavioral: Interaction Standard Theory-Based Multi-Care Program
- Conventional Nursing Intervention Group (Active Comparator): Participants received standard conventional nursing interventions as per the hospital's established protocol for postpartum hemorrhage management. This included careful examination of the soft birth canal and placenta, monitoring vital signs, administering oxygen therapy or blood transfusion if indicated, maintaining communication with the patient's family, and providing basic oral education regarding routine postpartum self-care.
  Interventions: Behavioral: Conventional Nursing Intervention

INTERVENTIONS:
Behavioral: Interaction Standard Theory-Based Multi-Care Program — A comprehensive nursing program based on King's Theory of Goal Attainment and Satir's model, focusing on structured nurse-patient communication, shared goal-setting, and multi-dimensional care addressing cognitive, psychological, behavioral, and dietary aspects. Delivered daily during hospitalization (30-45 min sessions) with post-discharge follow-up.
  Arms: Interaction Standard Theory-Based Multi-Care Program Group
Behavioral: Conventional Nursing Intervention — Standard hospital protocol for postpartum hemorrhage management including physiological monitoring, emergency measures as needed, and basic postpartum care education.
  Arms: Conventional Nursing Intervention Group

SUMMARY:
This study explored the impact of an interaction standard theory-based multi-care program on postpartum recovery, coping styles, psychological distress, and quality of life in women experiencing postpartum hemorrhage (PPH). A total of 110 women with PPH were randomized into a study group receiving the multi-care program or a control group receiving conventional nursing. Outcomes were assessed at baseline and 2 weeks post-intervention. The multi-care program significantly improved postpartum recovery, enhanced adaptive coping, reduced psychological distress, and improved quality of life compared to conventional care.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a severe obstetric complication. While standard medical care addresses the physiological crisis, the psychosocial needs and coping mechanisms of women experiencing PPH may be inadequately addressed by conventional nursing. This prospective, randomized controlled trial aimed to evaluate an interaction standard theory-based multi-care program, integrating King's Theory of Goal Attainment and Satir's model, for women with PPH. Participants (n=110) admitted to Shijiazhuang Obstetrics and Gynecology Hospital from October 2023 to October 2024 were randomly assigned to the study group (n=55) receiving the multi-care program or the control group (n=55) receiving conventional nursing. The multi-care program included collective training for nursing staff, individualized patient data collection, collaborative care plan development, and specific interventions in hemorrhage care, psychological care (empathetic listening, Satir's communication stances, music therapy, guided imagery), cognitive intervention (education on PPH), dietary care, and rehabilitation training. Follow-up occurred at 1 and 2 weeks post-discharge. The study assessed changes in coping styles (SCSQ), psychological distress (HAMD, HAMA), quality of life (WHOQOL-BREF), postpartum recovery indicators (lochia duration, lactation onset, uterine involution, hospital stay), and nursing satisfaction. The study was designed and reported following CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Delivered in our hospital and received postpartum treatment, with a blood loss >500 mL within 24 hours after delivery;
* Age <40 years;
* Single live birth at full term;
* Stable vital signs;
* No pregnancy-related complications (other than PPH itself post-diagnosis);
* Clear cognitive function and self-awareness;
* Normal hearing and communication ability.

Exclusion Criteria:

* Cervical laceration (as primary cause of PPH if not manageable by standard protocol and requiring extensive surgical repair beyond typical scope);
* Pre-existing severe cardiovascular diseases;
* Pre-existing severe renal, cardiac, or hepatic insufficiency;
* Known pre-existing coagulation disorders;
* Active systemic infectious diseases;
* Malignant tumors;
* Cellular immune function defects;
* Incomplete data or withdrawal from the study (prior to completion of the 2-week follow-up, though none occurred).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Coping Styles (Positive Coping) | Baseline (1 day post-PPH event) and 2 weeks post-intervention.
  Assessed using the Simplified Coping Style Questionnaire (SCSQ) positive coping subscale (0-36 points). Higher scores indicate more positive coping.
Change in Coping Styles (Negative Coping) | Baseline (1 day post-PPH event) and 2 weeks post-intervention.
  Assessed using the Simplified Coping Style Questionnaire (SCSQ) negative coping subscale (0-24 points). Lower scores indicate less negative coping.
Change in Depression Severity | Baseline (1 day post-PPH event) and 2 weeks post-intervention (or 1 day before discharge if earlier).
  Assessed using the Hamilton Depression Rating Scale (HAMD-17). Total score ranges, with scores >24 indicating severe depression, 18-24 moderate, 7-17 mild. Lower scores indicate less depression.
Change in Anxiety Severity | Baseline (1 day post-PPH event) and 2 weeks post-intervention (or 1 day before discharge if earlier).
  Assessed using the Hamilton Anxiety Rating Scale (HAMA). Total score up to 56, with scores ≥29 severe anxiety, ≥21 definite, ≥14 mild, ≥7 possible. Lower scores indicate less anxiety.
Change in Quality of Life | Baseline (1 day post-PPH event) and 2 weeks post-intervention.
  Assessed using the World Health Organization Quality of Life Brief Version (WHOQOL-BREF). Consists of 26 items across four dimensions (Environment, Physical, Psychological, Social Relations). Each item scored 0-5, higher total scores indicate better quality of life.
Duration of Lochia | Assessed up to 2 weeks post-intervention.
  Time in days from delivery until lochia cessation.
Time for Uterus to Return to Pelvic Cavity (Uterine Involution) | Assessed up to 2 weeks post-intervention.
  Time in days from delivery for the uterus to involute to the pelvic cavity.
Length of Hospitalization | From enrollment until hospital discharge (up to approximately 1 week)
  Duration of hospital stay in days post-PPH event.

SECONDARY OUTCOMES:
Nursing Satisfaction Rate | At discharge (within 2 weeks post-intervention).
  Assessed using a locally adapted patient satisfaction questionnaire (15 items) focusing on nursing care. Levels: satisfied, neutral, dissatisfied. Rate calculated as (Number of satisfied + neutral patients) / Total number of patients × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, Principal Investigator — Shijiazhuang Obstetrics and Gynecology Hospital
Locations (1):
- Shijiazhuang Obstetrics and Gynecology Hospital, Shijiazhuang, Hebei, China